CLINICAL TRIAL: NCT04211558
Title: A Phase 1, Open-Label Study to Evaluate the Pharmacokinetics of Single Oral Doses of Ozanimod in Healthy Adult Chinese Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics of Single Oral Doses of Ozanimod in Healthy Adult Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPC-1063-CP-002; U1111-1244-6464 (Other: WHO)
Record Dates: First submitted 2019-12-24; First posted 2019-12-26 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; Pharmacokinetics (PK); Ozanimod; Adult Chinese Subjects
MeSH Terms: interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozanimod 0.46mg (Experimental): Ozanimod single doses of 0.46 mg (1 x 0.46 mg capsule) will be administered on Day 1. Ozanimod will be administered following an overnight fast of at least 10 hours before dosing and with approximately 240 mL of nonrefrigerated, noncarbonated water (additional water may be allowed if required for the subject to complete dosing). Subjects will remain fasted for 4 hours after ozanimod dosing.
  Interventions: Drug: Ozanimod
- Ozanimod 0.92mg (Experimental): Ozanimod single doses of 0.92 mg (1 x 0.92-mg capsule) will be administered on Day 1. Ozanimod will be administered following an overnight fast of at least 10 hours before dosing and with approximately 240 mL of nonrefrigerated, noncarbonated water (additional water may be allowed if required for the subject to complete dosing). Subjects will remain fasted for 4 hours after ozanimod dosing.
  Interventions: Drug: Ozanimod

INTERVENTIONS:
Drug: Ozanimod — Ozanimod

SUMMARY:
This is a Phase 1, open-label, single-dose study. Approximately 24 Chinese healthy adult subjects will be enrolled to receive a single oral dose of ozanimod 0.46 mg or 0.92 mg (12 subjects per dose cohort).

Subjects will be screened for participation within 28 days prior to dosing. Eligible subjects will be admitted to the clinical research unit (CRU) or hospital one day before dosing (Day -1) and will be domiciled until Day 15 (approximately 336 hours after ozanimod dosing). Serial PK blood samples for the measurement of plasma concentrations of ozanimod and active metabolites will be collected predose and up to 336 hours after ozanimod dosing.

Physical examinations,12-lead electrocardiograms (ECGs) and ambulatory ECGs, vital sign measurements,pulmonary function tests (PFTs), and clinical laboratory tests will be performed and adverse events and concomitant medications will be monitored throughout the study to assess safety.

Subjects will be contacted by telephone approximately 30 ± 5 days after dosing for a follow-up safety assessment.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is a male or female, ages 18 to 45 years
2. Subject is of Chinese origin; individual currently residing in mainland China who was born in China and has both parents of Chinese descent
3. Female subjects must meet at least 1 of the following criteria:

   * Negative serum pregnancy test at Screening and Day -1
   * Postmenopausal
   * Received surgical sterilization at least 6 months before Screening with medical records.
4. Females of child-bearing potential:

   Must agree to practice a highly effective method of contraception throughout the study until 90 days postdose. Highly effective methods of contraception are those that alone or in combination result in a failure rate of a Pearl index of less than 1% per year when used consistently and correctly.

   All subjects:

   Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception.
5. Subject has a total body weight of at least 50 kg (110 lbs); body mass index (BMI) within the range of 19.0 to 24.0 kg/m2
6. Subject is in good health, as determined by no clinically significant findings from medical or surgical history, 12-lead ECG, physical examination, clinical laboratory tests, and vital signs.
7. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
8. Subject is willing and able to adhere to the study visit schedule and other protocol

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject with a seated blood pressure outside 90 to 140 mmHg systolic or 50 to 90 mmHg diastolic at Screening or Day -1.
2. Subject with a seated pulse rate outside 55 to 90 bpm at Screening or Day -1.
3. Subject has a presence or history of any abnormality or illness that, in the opinion of the Investigator, may affect absorption, distribution, metabolism, or elimination of the IP(s) or would limit the subject's ability to participate in and complete this clinical study.
4. Subject has a history of alcoholism, drug abuse, or addiction within 24 months prior to Screening.
5. Subject has a positive serum test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
6. Subject has used any tobacco- or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, electronic cigarettes, vape, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) or marijuana (cigarette, joint, vape, edibles, etc) within 3 months prior to dosing of the IP.
7. Subject has a positive urine drug test including cotinine at Screening or Day -1.
8. Subject has a positive alcohol urine or breath test at Screening or Day -1.
9. Subject has received any investigational drug within 30 days or 5 times the elimination half-life (if known), whichever is longer, prior to dosing of the IP.
10. Subject has used any systemic over-the-counter medication (excluding acetaminophen up to 1 g/day), dietary or herbal supplement including traditional Chinese medicine (excluding vitamins/multivitamins) within 14 days prior to the first dose of IP. St. John's wort, naringenin, curcumin/turmeric, passion flower, and quercetin must be discontinued at least 28 days prior to dosing of the IP.
11. Subject has used any systemic prescription medication (excluding hormonal contraceptives) within 28 days or 5 times the elimination half-life, whichever is longer, prior to dosing of the IP.
12. Subject has ingested alcohol within 7 days prior to dosing of the IP.
13. Subject fails or is unwilling to abstain from strenuous physical activities for at least 24 hours prior to dosing of the IP.
14. Subject has poor peripheral venous access.
15. Subject has donated greater than 400 mL of blood within 60 days prior to dosing of the IP or the subject has accepted a blood transfusion or received blood products.
16. Subject has had surgery within 4 weeks prior to dosing, or plans to have surgery during the study period.
17. Subject has a special diet requirement and cannot follow the CRU's or hospital's standard meal.
18. Subject drink large amounts of tea, coffee and or caffeinated drinks (>8 cups/day, 1 cup = 250mL) daily.
19. Subject has a history of any medical condition or medical history that, in the opinion of the Investigator, might confound the results of the study or jeopardize the safety or welfare of the subject.
20. Subject has history of hypersensitivity or allergic reaction to food or other drugs including S1P receptor modulators.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic - Cmax (Ozanimod, CC112273 and CC1084037) | 14 days
  Maximum observed plasma concentration within the dosing interval
Pharmacokinetic - Tmax (Ozanimod, CC112273 and CC1084037) | 14 days
  Time to Cmax
Pharmacokinetic - AUC∞ (Ozanimod) | 14 days
  Area under the concentration-time curve from time 0 to infinity
Pharmacokinetic - CL/F (Ozanimod) | 14 days
  Apparent oral clearance
Pharmacokinetic - Vz/F (Ozanimod) | 14 days
  Apparent volume of distribution during terminal phase after oral administration
Pharmacokinetic - t1/2 (Ozanimod, CC112273 and CC1084037) | 14 days
  Terminal elimination half-life
Pharmacokinetic - AUClast (CC112273 and CC1084037) | 14 days
  Area under the concentration-time curve from time 0 to time of last quantifiable concentration
Pharmacokinetic - AUC0-14d (CC112273 and CC1084037) | 14 days
  Area under the concentration-time curve from time 0 to 14 days postdose

SECONDARY OUTCOMES:
Adverse Events (AEs) | From consent until 30 days after the last dose of IP
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a pre-existing condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Peijin Zhang, M.D, PhD, Study Director — Bristol-Myers Squibb
Locations (1):
- Capital Medical University - Beijing Anzhen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/